CLINICAL TRIAL: NCT02044146
Title: Reassessment of Anti-Platelet Therapy Using InDividualized Strategies - Modifying Acute CoroNary Syndrome Algorithms Based on Genetic and Demographic Evaluation: The RAPID-MANAGE Study
Brief Title: A Pharmacodynamic Study of a Personalized Strategy for P2Y12 Inhibition Versus Ticagrelor in Reducing Ischemic and Bleeding Risk
Acronym: RAPID MANAGE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Derek So, Associate Professor, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20130601
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Personalized Therapy (Experimental): A point-of-care bedside genetic test for CYP2C19*2 and CYP2C19*3 using a buccal swab will be conducted.2 P2Y12 inhibitory drug therapy will be then be directed based on a risk algorithm (integrating genotyping and clinical variables). Patients with "high ischemic risk" are defined as having (*2 or *3) and/or diabetes and/or (having age>65 AND BMI>=28). "High-risk" patients will be switched to prasugrel at 10mg daily, while "low ischemic risk" patients be kept on clopidogrel 75 daily. For patients >age 75 or wt < 60 kg, prasugrel will be reduced to 5mg daily.
  Interventions: Drug: Ticagrelor, Prasugrel, Clopidogrel
- Ticagrelor (Active Comparator): Patients will be treated with a 90mg twice daily regimen of Ticagrelor
  Interventions: Drug: Ticagrelor, Prasugrel, Clopidogrel
- Clopidogrel registry arm (Other): A concurrent registry of patients (not randomized) who are receiving clopidogrel only (as decided by treating physician) will be followed as a comparator group.
  Interventions: Drug: Ticagrelor, Prasugrel, Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor, Prasugrel, Clopidogrel

SUMMARY:
In patients with heart attacks, the treatment of choice is to restore blood flow with percutaneous coronary intervention (PCI) (use of stents (metal meshes) to open blockages). After PCI, the standard drug treatment includes aspirin and clopidogrel. These medications block full function of the platelet cells, which are responsible for clotting. Despite their use, patients after PCI are at risk for heart attacks, sudden clotting of stents or death. A major contributor may be resistance to clopidogrel. New more potent drugs, which can overcome the resistance, are now available; however, they come with an increase chance of severe bleeding and costs. An ideal solution would be to identify at-risk patients and selectively treat them with more potent drugs, while lower-risk patients continue with clopidogrel. This type of strategy (personalized strategy) would decrease heart attacks and death (compared to clopidogrel), while also preventing bleeding complications (compared to treating all patients with the new drugs).

Of resistant patients, many carry genes (inherited units) that prevent proper absorption of clopidogrel. Our group has developed and tested a new bedside genetic test, which identifies carriers of at-risk genes. However, this technique alone does not identify all at-risk patients. Consequently, we have now devised a novel tool, which combines genetics with patient characteristics to identify high-risk patients.

The present study combines this new tool into a strategy for personalized treatment. Patients with heart attacks who undergo PCI will be randomly assigned to 1 of 3 strategies: a) new personalized strategy, b) clopidogrel strategy (previous standard drug) or c) ticagrelor strategy (stronger approved drug). The function of the platelet cells will be measured at 1 month to determine potential benefits. Evaluation of this new personalized strategy is important for improving patient outcomes after PCI. The hypothesis is that patients receiving a personalized strategy will have decrease risk for future heart attacks and bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients: age >18 yrs, < 75yrs

  -> 60 kg ( since March 2015 age >75 and < 60 kg eligible - but prasugrel reduced to 5mg daily if randomized to personalized therapy arm)
* NSTEMI undergoing PCI will be eligible

Exclusion Criteria:

- Patients will be excluded if they have: i) a contra-indication for clopidogrel or prasugrel or ticagrelor (as per monograph), ii) have an intolerance to aspirin, iii) have absolute requirement for ticagrelor or prasugrel (e.g. stent thrombosis, allergic reaction to clopidogrel), iv) requirement for anti-coagulation treatment, v) a history of stroke, TIA or intracranial hemorrhage , vi) a platelet count < 100,000/μl, vii) a known bleeding diathesis, viii) hematocrit <30% or >52%, ix) severe liver dysfunction, x) renal insufficiency (creatinine clearance < 30ml/min), xi) adjuvant therapy with a glycoprotein IIbIIIa inhibitor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients in Therapeutic Window | 1 month
  The primary endpoint is the proportion of patients outside of the "therapeutic window" in the personalized therapy (PN) arm compared to the ticagrelor (TG) arm at 1 month. The "therapeutic window" will be defined by platelet function values (VerifyNow P2Y12 assay - P2Y12 reaction unit (PRU) ≤ 208 (correlated with decreased ischemic outcomes) AND PRU >= 85 (correlated with decrease bleeding). This is a surrogate of NACE (net adverse clinical events)

SECONDARY OUTCOMES:
P2Y12 Reaction Unit (PRU) | Baseline, Day 1, 1 month
  change in PRU from baseline, day 1 to 1 month in each of the groups
Bleeding | 1 month, 6 months
  the incidence of bleeding (defined by TIMI minor and major bleeds) among groups
MACE | 1 month, 6 months
  combined clinical endpoint (MACE) including death, myocardial infarction(MI) or urgent target vessel revascularization (TVR)
Stent thrombosis | 1 month, 6 month
  stent thrombosis (ARC definite/probable)

OTHER OUTCOMES:
Cost | 1 month, 6 months
  Evaluate cost involved in each strategy
Genetic factors associated to outcomes | 1 month, 6 months
  Exploratory analysis of other potential genetic variants to outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec